CLINICAL TRIAL: NCT02981836
Title: A Blind, Randomized and Controlled Clinical Trial to Evaluate the Protective Effect, Safety and Immunogenicity of Live Attenuated Varicella Vaccines for Healthy Children
Brief Title: A Blind, Randomized and Controlled Study of Live Attenuated Varicella Vaccines
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Sinovac (Dalian) Vaccine Technology Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: PRO-VZV-3001
Record Dates: First submitted 2016-11-28; First posted 2016-12-05 (Estimated); Last update posted 2017-10-26 (Actual); Status verified 2016-11

CONDITIONS: Varicella
Keywords: live attenuated varicella vaccine; protective effect; safety; immunogenicity; child
MeSH Terms: conditions — Chickenpox

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Experimental Group (Experimental): * Single intramuscular injection of the investigational vaccine (0.5 ml) on Day 0;
  * Intervention: investigational live attenuated varicella vaccine;
  Interventions: Biological: Investigational live attenuated varicella vaccine
- Control Group (Sham Comparator): * Single intramuscular injection of the diluent of lyophilized vaccine (0.5 ml) on Day 0;
  * Intervention: diluent of lyophilized vaccine;
  Interventions: Biological: diluent of lyophilized vaccine

INTERVENTIONS:
Biological: Investigational live attenuated varicella vaccine — The investigational vaccine was manufactured by Sinovac (Dalian) Vaccine Technology Co., Ltd.
  Arms: Experimental Group
Biological: diluent of lyophilized vaccine — The diluent of lyophilized vaccine was manufactured by Sinovac (Dalian) Vaccine Technology Co., Ltd.
  Arms: Control Group

SUMMARY:
The purpose of this study is to evaluate the protective effect, safety and immunogenicity of a live attenuated varicella vaccine in healthy children.

DETAILED DESCRIPTION:
This study is a randomized, blind, controlled phase III clinical trial. The purpose of this study is to evaluate the protective effect, safety and immunogenicity of a live attenuated varicella vaccine manufactured by Sinovac (Dalian) Vaccine Technology Co., Ltd. The control is diluent of lyophilized vaccine manufactured by Sinovac (Dalian) Vaccine Technology Co., Ltd. All participants are healthy, and will be randomly assigned into experimental group or control group in the ratio 1:1.

ELIGIBILITY:
Inclusion Criteria:

* Healthy volunteer between 1 - 12 years old;
* Proven legal identity;
* Guardian(s) of the volunteer and/or volunteers themselves should be capable of understanding the written consent form, and such form should be signed before the volunteer being included into this study;

Exclusion Criteria:

* Prior vaccination with varicella vaccine or with history of varicella zoster virus (VZV) infection;
* Axillaty temperature > 37.0 °C;
* History of allergy to any vaccine or vaccine ingredient, or serious adverse reaction(s) to vaccination, such as urticaria, difficulty in breathing, angioneurotic edema, abdominal pain, etc;
* History of epilepsy, seizures or convulsions, or a family history of mental illness, autoimmune disease or immunodeficiency;
* Severe malnutrition, congenital malformation, developmental disorders, or serious chronic diseases;
* Acute disease or acute stage of chronic disease within 7 days prior to study entry;
* Receipt of any of the following products:

  1. Any subunit vaccine or inactivated vaccine within 7 days prior to study entry;
  2. Any live attenuated vaccine within 1 month prior to study entry;
  3. Any blood product, immunosuppressant, hormone, or other investigational medicine(s) within 30 days prior to study entry;
* Any significant abnormity of heart, lung, skin, or pharynx;
* Any other factor that suggesting the volunteer is unsuitable for this study based on the opinions of investigators;

Ages: 1 Year to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 5997 (Actual)
Dates: Start 2016-08 (Actual); Primary Completion 2017-06 (Actual); Study Completion 2017-09 (Actual)

PRIMARY OUTCOMES:
The incidences of varicella of each group | ≥30 cases reported 30 days after injection
  The first 30 cases of varicella occurred 30 days after injection will be collected.
The protection rate of the vaccine | ≥30 cases reported after 30 days of the injection
  The protection rate will be calculated based on the reported cases occurred 30 days after injection.

SECONDARY OUTCOMES:
The incidences of adverse events (AEs) of each group | 30 days
  AEs occurred within 30 days after injection will be collected.
The incidences of serious adverse events (SAEs) of each group | 6 months
  SAEs occurred within 6 months after injection will be collected.
The seroconversion rate of the immunogenicity group | 30 days after injection
  Seroconversion rate of the immonogenicity group 30 days after injection will be collected.
The geometric mean titer (GMT) of the immunogenicity group | 30 days
  Geometric mean titer (GMT) of the immonogenicity group will be collected before and 30 days after injection.
The geometric mean fold increase (GMI) of the immunogenicity group | 30 days after injection
  Geometric mean fold increse (GMI) of the immonogenicity group will be calculated based on the geometric mean titer.

CONTACTS AND LOCATIONS:
Overall Officials: Shengli Xia, Principal Investigator — Henan Provincial Center for Disease Control and Prevention
Locations (2):
- China (2):
  - Xiangcheng County Center for Disease Control and Prevention, Xuchang, Henan
  - Biyang County Center for Disease Control and Prevention, Zhumadian, Henan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Zhang Y, Wang L, Wang Y, Zhang W, Jia N, Xie Z, Huang L, You W, Lu W, Li E, Gao F, Hu Y, Meng F, Xia S. Immunogenicity and Safety of a Booster Dose of Live Attenuated Varicella Vaccine, and Immune Persistence of a Primary Dose for Children Aged 2 to 6 Years. Vaccines (Basel). 2022 Apr 22;10(5):660. doi: 10.3390/vaccines10050660. PMID 35632416
- [Derived] Hao B, Chen Z, Zeng G, Huang L, Luan C, Xie Z, Chen J, Bao M, Tian X, Xu B, Wang Y, Wu J, Xia S, Yuan L, Huang J. Efficacy, safety and immunogenicity of live attenuated varicella vaccine in healthy children in China: double-blind, randomized, placebo-controlled clinical trial. Clin Microbiol Infect. 2019 Aug;25(8):1026-1031. doi: 10.1016/j.cmi.2018.12.033. Epub 2019 Jan 4. PMID 30616012